CLINICAL TRIAL: NCT00340561
Title: Effects of Experience on the Driving Performance of Novice Teen Drivers
Brief Title: Effect of Experience on Driving Performance in New Teenage Drivers
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905070; 05-CH-N070
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-07

CONDITIONS: Learning
Keywords: Test Track; Distraction; Motor Vehicle; Learning; Inexperience

SUMMARY:
This study will evaluate the driving performance of new teenage drivers and determine to what extent independent driving experience improves driving performance of young drivers. Motor vehicle crash rates are highest among new teen drivers, especially during the first 6 months and 1,000 miles of independent licensed driving. Crash rates decline with experience, and this study will assess the effect of driving experience on performance.

Newly licensed teenagers ranging from 16 years, 3 months to 17 years of age and experienced drivers 30 to 50 years of age may be eligible for this study. Candidates must be able to legally drive in the commonwealth of Virginia and have at least 20/40 correctable vision.

Participants complete a questionnaire about their health and driving experience. They are then tested on a driving test track. Teens are tested within 3 weeks of obtaining their driver's license and before they have more than 100 miles of independent driving experience. They are tested a second time 6 to 12 months later and after they have more than 1,000 miles of driving experience. A group of experienced adult drivers are also tested to provide a comparison.

The driving test is conducted on a smart road - a controlled, 2.2-mile two-lane research track at the Virginia Tech Transportation Institute. It is designed for safety, with restricted access, nothing for a vehicle to hit, carefully placed guardrails, and other safety features. The research vehicle is equipped with airbags, anti-lock brakes, and other safety equipment. It also has sensors and tiny video cameras to assess the behavior of the vehicle and the driver; this equipment does not interfere with the operation of the vehicle.

An experimenter accompanies the driver and instructs him or her to perform routine driving skills, such as stopping, changing lanes and maintaining speed, as well as to other tasks such as inserting a CD into an entertainment console, having a conversation, and answering a cellular telephone call. The driver has an opportunity to practice the tasks before being tested.

The driver's speed is limited to 35 mph or less during the experiment and the driver is required to wear seat belts and follow safe driving procedures. The experimenter is in the front passenger seat can stop the vehicle using a separate brake pedal.

DETAILED DESCRIPTION:
Motor vehicle crash rates are highest among novice teen drivers, especially during the first six months and 1000 miles of independent licensed driving. Crash rates decline with driving experience, however, no research has demonstrated learning effects on performance due to independent driving experience and the extent and variability in driving performance among novice young drivers has not been established. The purpose of this study is to assess the effect of driving experience on driving performance. We propose to use standard measures of driving performance under controlled experimental conditions on a driving test-track and vehicle designed for this purpose. Specifically, we propose to test the driving performance of a sample of teens within a few weeks after licensure while they are still relatively inexperienced drivers and again after greater than 6 months and 1000 miles of driving experience test their driving performance. A sample of experience adult drivers would be tested in similar fashion to provide an additional comparison group.

ELIGIBILITY:
* INCLUSION CRITERIA:

Recruitment of teen participants will occur by arrangement with local driving schools in Montgomery County, VA.

Potential participants aged 16 or 17 who have held their driver's license for one month or less may be eligible.

Participants may be recruited during their training, and will only be eligible after they have met all requirements for licensure, and after both parental consent and teen assent are obtained.

If the teen wishes to participate, they must have their parent or legal guardian speak to the VTTI experimenter over the telephone for screening and then accompany the teen at an appointment so that the study can be explained and consent and assent provided.

Experienced adult drivers will be recruited via one-page recruitment fliers describing the study posted in the Blacksburg, VA area.

After an appointment is made, a telephone screening will occur using the Telephone Driver Screening and Demographic Questionnaire to assess age, sex, medical and driving history.

Ages: 7 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48
Dates: Start 2005-01; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Doherty ST, Andrey JC, MacGregor C. The situational risks of young drivers: the influence of passengers, time of day and day of week on accident rates. Accid Anal Prev. 1998 Jan;30(1):45-52. doi: 10.1016/s0001-4575(97)00060-2. PMID 9542543